CLINICAL TRIAL: NCT07152340
Title: The Safety and Efficacy of Sequential Hormone Therapy and IBI311 Therapy in Patients With Active Moderate to Severe TAO in the Initial Treatment.
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Changzheng Hospital (Other)
Responsible Party: Principal Investigator, Tuo Li, MD, Deputy Director, Shanghai Changzheng Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASAP-1
Record Dates: First submitted 2025-06-14; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-06

CONDITIONS: Thyroid Associated Ophthalmopathies
Keywords: IGF-1R; TED; glucocorticoids; MRI imaging
MeSH Terms: conditions — Graves Ophthalmopathy; Insulin-Like Growth Factor I, Resistance To | interventions — Glucocorticoids

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IBI311 (Active Comparator): 8 infusions of teprotumumab (10 mg/kg for the first infusion and 20 mg/kg for the remaining 7 infusions)
  Interventions: Drug: IBI311
- Glucocorticoid (Active Comparator): Patients with active thyroid ophthalmopathy will receive 500 mg of methylprednasone intravenous injection once a day for 3 days, followed by once every 2 weeks, for a total of 8 times.
  Interventions: Drug: Glucocorticoids

INTERVENTIONS:
Drug: IBI311 — IBI311 is a fully human anti-IGF-1R mAb. IBI311 will be provided in single-dose 10-mL glass vials as a Injection solution containing.
  Arms: IBI311
Drug: Glucocorticoids — 500mg methylprednisolone was intravenously injected once a day for 3 consecutive days. The next treatment was carried out with an interval of 2 weeks for a total of 8 times.
  Arms: Glucocorticoid

SUMMARY:
Thyroid-associated ophthalmopathy (TAO) is an organ-specific autoimmune disease closely related to thyroid disease, which leads the incidence of orbital disease in adults and is the most common cause of diffuse toxic goiter (Graves disease, GD). The clinical manifestations of TAO are complex and varied. In severe cases, it may seriously impair visual function, affect daily life, and even cause corneal ulceration, perforation, and blindness. Therefore, a reasonable and effective treatment plan should be chosen according to the degree of TAO.

Tetuzumab (IBI311) is a fully human monoclonal insulin-like growth factor-1 receptor inhibitory antibody. It has binding activity against IGF-1R positive cells, can block the binding of IGF-1 and IGF-2 to IGF-1R, and has a dose-dependent effect. It can inhibit the proliferation of HT29 cells caused by the activation of the IGF-1R signaling pathway. Meanwhile, it can dose-dependently inhibit the proliferation of orbital fibroblasts and the secretion of hyaluronic acid (HA) in patients with TAO.

However, there are still significant gaps in the existing research evidence: the lack of head-to-head studies of temumab and glucocorticoids.

The aim of this clinical study is to:

1. To evaluate the efficacy of IBI311 treatment in patients with active moderate to severe TAO in the initial treatment.
2. To observe the safety of IBI311 treatment in patients with active moderate to severe TAO in the initial treatment.
3. Head-to-head comparison of sequential hormone therapy and IBI311 therapy in patients with active moderate to severe TAO in the initial treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with TAO by Bartley criteria.
* Moderate to severe patients defined by EUGOGO.
* CAS ≥4 (on the 7-item scale) for the study eye.
* Have not received glucocorticoid treatment for TAO in the past.

Exclusion Criteria:

* Anticipated need for intervention due to sight-threatening complications or other significant and acute deterioration in vision.
* Combined with other lesions in the orbit.
* Receive orbital radiotherapy or surgical treatment for TED, including orbital decompression, strabismus surgery and eyelid retraction correction.
* During the screening period, if either ear has a history of tinnitus or other hearing impairment; Or abnormal pure tone audiometry results (defined as an average bone conduction hearing threshold of ≥25 dB at 0.5, 1, 2, 4 kHz or a bone conduction hearing threshold of ≥40 dB at any frequency).
* At the time of screening, aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 3 times ULN, or accompanied by active hepatitis B (defined as HBsAg positive with HBV-DNA load greater than 1000 IU/mL), or being receiving anti-hepatitis B virus treatment.
* During screening, the Glomerular Filtration Rate (GFR) was < 30 ml/min/1.73m2 (using the MDRD formula: GFR =186× serum creatinine (mg/dl) -1.154× (age) -0.203× (0.742 [if female]), unit conversion of serum creatinine: 1 μmol/L=0.0113 mg/dL); 10) At the time of screening, there was poorly controlled diabetes (defined as glycated hemoglobin ≥7.0% at the time of screening, or a new diabetes drug [oral or injection] or a dose change of the current prescribed diabetes drug > 10% within 60 days before screening).
* Screening for poorly controlled hypertension, with systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥100 mmHg; Or adjust the antihypertensive drug (dosage or type of drug) within 30 days before screening; Evidence of renal artery stenosis or unstable blood pressure (including orthostatic hypotension, etc.).
* At the time of screening, the 12-lead ECG showed a heart rate of < 50 beats/min or > 100 beats/min. The ECG indicated active heart disease, or the researchers believed that the abnormal ECG at the time of screening would interfere with the interpretation of the ECG results in the subsequent follow-up process. Especially, QTcF > 450 ms (for men) and QTcF > 470 ms (for women) should be excluded.
* HIV antibody or HCV antibody positive individuals or those with active syphilis (defined as those with positive non-specific syphilis antibodies or those who need anti-syphilis treatment after consultation by the infectious disease department).
* History of systemic (eg, oral or IV) steroid use of methylprednisolone for the treatment of TAO.
* Any major illness/condition or evidence of an unstable clinical condition that, in the investigators judgment, will substantially increase the risk to the participant, or confound the interpretation of safety assessments, if they were to participate in the study.
* Any other condition that, in the opinion of the investigator, would impair the ability of the participant to comply with the study procedures or impair the ability to interpret data from the participants participation in the study.
* Pregnant or lactating.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2030-05-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants who were overall treatment responders ater 4 times and at the end of treatment | up to 24 weeks
  Subjects in the study eye with a reduction of ≥2 mm in exophthalmos and a reduction of ≥2 points in the clinical activity score (CAS) from baseline, and no deterioration in the contralateral eye (an increase of ≥2 mm in exophthalmos or an increase of ≥2 points in CAS)
Percentage of participants who were CAS categorical responders after 4 times and at the end of the treatment | up to 24 weeks
  The CAS is a 7-item description of clinical activity, including:
  1. Spontaneous orbital pain;
  2. Gaze evoked orbital pain;
  3. Eyelid swelling that is considered to be due to active (inflammatory phase) thyroid eye disease/ Graves' Ophthalmopathy or Orbitopathy (TED/GO);
  4. Eyelid erythema;
  5. Conjunctival redness that is considered to be due to active (inflammatory phase) TED/GO (ignore "equivocal" redness);
  6. Chemosis;
  7. Inflammation of caruncle or plica. Each item is scored (1=present; 0=absent) and scores for each item are summed for total score of 0 (no inflammatory symptoms) to 7 (most inflammatory symptoms).
  CAS categorical responders were defined as subjects whose CAS in the study eyes decreased to 0 or 1 (with no or minimal inflammatory symptoms)
Percentage of participants who were diplopia responders after 4 times and at the end of the treatment | up to 24 weeks
  Diplopia responders were defined as percentage of participants with ≥ 1 class improvement of eye motility from baseline assessed by Gorman score.
  Gorman score: 1 = no diplopia, 2 =intermittent diplopia, 3 = inconstant (gaze-evoked) diplopia, 4 = constant diplopia in primary or reading position.
Percentage of participants who were proptosis responders after 4 times and and the end of the treatment | up to 24 weeks
  Proptosis responders were defined as subjects whose exophthalmos in the study eye decreased by ≥2 mm compared to the baseline, and whose exophthalmos in the contralateral eye did not deteriorate (increase by ≥2 mm) at the end of the intervention observation period -1.
Percentage of participants who were ATA categorical responders after 4 times and at the end of the treatment | up to 24 weeks
  Participants whose baseline ATA score of the study eye was >4, with a reduction of ≥1 grade in the ATA score, while there was no corresponding deterioration in the contralateral eye (≥1 grade deterioration).
  The denominator is the number of subjects with a baseline ATA score grade >4.

SECONDARY OUTCOMES:
Incidence and characterization of nonserious treatment emergent adverse events (TEAEs) during the treatment | through study completion, an average of 1 year
change of GO-QoL from baseline after 4 times and at the end of the treatment | up to 24 weeks
Changes of the visual field in the dark areas from baseline after 4 times and at the end of the treatment | up to 24 weeks

OTHER OUTCOMES:
MR Imaging changes of orbital contents compared with the baseline after 4 times and at the end of the treatment | up to 24 weeks
  Including: exophthalmos, the volume of the lacrimal gland/optic nerve/extraocular muscle/retroorbital adipose tissue/lacrimal gland, edema, inflammation, blood perfusion, fibrosis, and fatty changes

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Shanghai Changzheng Hospital, Changhua, Shanghai Municipality
  - Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Undecided